CLINICAL TRIAL: NCT07206134
Title: Modified Omega Bone Plate Versus Conventional Miniplates for Fixation of Mandibular Fractures in Mental Nerve Region
Brief Title: Evaluation of Modified Omega Plate in the Management of Mandibular Fractures Compared With Conventional Fixation
Acronym: COMET-OMF
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Tanta University (Other)
Responsible Party: Principal Investigator, Mohamed sobhie abdelhameed, Principal Investigator, Teaching Assistant of Oral and Maxillofacial Surgery, Faculty of Dentistry, Tanta University, Tanta University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: TantaOMS-OMEGAvsCONV-2025
Record Dates: First submitted 2025-09-12; First posted 2025-10-03 (Actual); Last update posted 2025-10-03 (Actual); Status verified 2025-09

CONDITIONS: Mandibular Fractures; Fracture in Mental Nerve Region
MeSH Terms: conditions — Mandibular Fractures

STUDY DESIGN:
Intervention Model Description: Parallel assignment
Who Masked: Participant, Outcomes Assessor
Masking Description: using closed envelop for participants the data will be given to outcomes assessors without defining the intervention for each group
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Modified Omega bone plate used for fixation of mandibular fractures in mental foramen region (Experimental): Reflection of vestibular flap without dissection around mental bundle and fracture reduction and fixation with 3D Modified Omega bone plate
  Interventions: Procedure: Modified Omega bone plate for fixation of mandibular fractures in mental foramen region
- Conventional miniplates used for fixation of mandibular fractures in mental foramen region (Experimental): Reflection of vestibular flap and dissection around mental bundle and fracture reduction and fixation with 2 miniplates
  Interventions: Procedure: Conventional miniplates for fixation of mandibular fractures

INTERVENTIONS:
Procedure: Modified Omega bone plate for fixation of mandibular fractures in mental foramen region — Reflection of vestibular flap without dissection around mental bundle and fracture reduction and fixation with 3D Modified Omega bone plate
  Arms: Modified Omega bone plate used for fixation of mandibular fractures in mental foramen region
Procedure: Conventional miniplates for fixation of mandibular fractures — Reflection of vestibular flap with dissection around mental bundle and fracture reduction and fixation with 2 miniplates
  Arms: Conventional miniplates used for fixation of mandibular fractures in mental foramen region

SUMMARY:
Twelve adult patients with mandibular fractures in the mental region were enrolled and randomly divided into two equal groups. Group I received fixation using custom-designed modified omega bone plates, while Group II was treated with conventional titanium miniplates following Champy's technique. Virtual surgical planning and 3D printing technology were used to fabricate customized plates in Group I. Clinical and radiographic assessments were conducted immediately, at 1 week, 3 months, and 6 months postoperatively. Parameters evaluated included soft tissue healing, pain, facial edema, lower lip paresthesia, maximal mouth opening, occlusion, fracture stability, and hardware integrity.

DETAILED DESCRIPTION:
This study was conducted on twelve adult patients with mandibular fracture in mental nerve region, selected from the outpatient clinic, Oral and Maxillofacial Surgery Department, Faculty of Dentistry, Tanta University.

The selected patients were randomly divided into two equal groups, group I (6 patients) were treated by modified omega bone plate, while group II (6 patients) were treated by 2.0 mm conventional miniplates according to Champy's principle. A comparison between the two groups was conducted.

Modified Omega bone plate is a specially-designed, 8-hole, titanium miniplate modified by adding upper struts to the Ω symbol. It has lower horizontal struts (which provides stability along the lower border) with four holes, the proximal 2 holes are round and the distal are pear shape (compression holes). Two vertical struts at the ends of the horizontal struts (which provide resistance against the torsional forces),Upper horizontal struts (which counteract the tensional forces along the alveolar border) with four holes the proximal 2 holes are round and the distal are pear shape. The omega shape of this plate helps it to adapt easily around the mental neurovascular bundle.

Preoperative evaluation of the patients was carried out by taking history and performing clinical and radiographic examinations. Clinical examination included intraoral and extraoral inspection and palpation of the fracture sites. Radiographic examination was used to determine the site, number, type of fractures and degree of displacement.

Under general anesthesia, the fracture line was exposed through an intraoral approach, and the fracture segments were reduced. In group I, fixation of the reduced segments was done with modified omega bone plate which predetermined virtually. In group II, 2conventional miniplates placed on inferior border & subapical were used to fix the fracture.

Postoperative clinical evaluation were performed immediately, one week, two weeks, one month, three months and postoperative radiographic evaluation were performed immediately, three months and six months. The postoperative clinical evaluation included presence or absence of infection, bony union or stability, state of occlusion, maximal mouth opening, sensory nerve function, condition of teeth related to the fracture line and, patient's tolerance to the plate.

ELIGIBILITY:
Inclusion Criteria:

Patients with displaced mandibular parasymphysis or body fracture in the mental nerve region

Indicated for open reduction and internal fixation (ORIF)

Exclusion Criteria:

* Patients with systemic diseases that affect bone healing
* Fractures with crushed mental foramen
* Comminuted fractures where fixation is difficult
* Patients with anatomical variations (e.g., bifid inferior alveolar or mental nerve), based on preoperative CT nerve tracing

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2023-03-01 (Actual); Primary Completion 2024-12-01 (Actual); Study Completion 2025-08-04 (Actual)

PRIMARY OUTCOMES:
Pain intensity measured using Visual Analogue Scale (VAS) | At 1 day, 3 days, 1 week, and 1 month postoperatively
  Pain will be assessed using a 10-cm Visual Analogue Scale (VAS) ranging from 0 (no pain) to 10 (worst imaginable pain).

SECONDARY OUTCOMES:
Facial edema measured using linear facial measurements | At 1 day, 3 days, 1 week
  Edema will be assessed utilizing a horizontal and vertical guide with a tape on four reference points: outer canthus of the eye, angle of the mandible, tragus of the ear and outer corner of the mouth respectively. To obtain the percentage of facial swelling, the difference between measurements of the postoperative and preoperative periods will be divided by the value of the preoperative period.
  Souza JA, Consone DP. Method for measurement of facial edema after oral surgery.
Neurosensory function assessed by two point discrimination test | Up to 3 months
  Sensory function tested using caliber
Maximal Interincisal Opening (MIO) | Preoperative, and postoperative day 1, day 3, 1 week, and 1 month
  Measured using digital caliper between maxillary and mandibular central incisors.
Occlusion Status | Postoperative 1 week and 1 month
  Clinical evaluation of occlusion compared with pre-injury status using ulgics questionnaire
Operation Time | Intraoperative
  Total duration of surgery measured from first incision to last suture.
Interfragmentary Gap | 1 day Postoperative
  Linear measurement radiographically on immediate postoperative CT

CONTACTS AND LOCATIONS:
Locations (1):
- Egypt faculty of dentistry, tanta university, Tanta, Egypt